CLINICAL TRIAL: NCT06802822
Title: The PART PILOT STUDY: a Pilot Study to Inform the Feasibility of a Definitive Prospective Interventional Study to Prevent Allosensitization in Patients Who Have Failed a First Renal Transplant
Brief Title: Prevent Allosensitization in Patients Who Have Failed a First Renal Transplant (PART)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, John Gill, Transplant Nephrologist, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H24-02541
Record Dates: First submitted 2025-01-24; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Kidney Transplant; Kidney Transplant Failure; Immunosuppresion
Keywords: kidney transplant; kidney transplant failure; immunosuppression; sensitization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Patients will withdraw from immunosuppressant after 6 months post dialysis initiation
  Interventions: Drug: Prevention of Allosensitization
- Arm 2 (Active Comparator): Patients will withdraw from immunosuppressant after 24 months post dialysis initiation
  Interventions: Drug: Prevention of Allosensitization

INTERVENTIONS:
Drug: Prevention of Allosensitization — This study evaluates the impact of two different durations of immunosuppressive therapy on kidney transplant patients who return to dialysis after a failed transplant. One group will continue immunosuppressive therapy for two years, while the other will stop the therapy six months after starting dialysis. The goal is to determine if continuing immunosuppression can reduce the risk of allosensitization and improve outcomes, compared to stopping the therapy earlier.

SUMMARY:
Kidney transplant is often the best treatment for people with kidney failure, but transplanted kidneys don't always last a lifetime. Many transplanted kidneys fail within 12 years, leaving patients needing dialysis or another transplant. One major issue is something called "allosensitization," which happens when the immune system attacks the donated kidney due to foreign markers on the kidney. This makes it harder to match a patient with another donor kidney in the future.

To try to prevent this, patients are given immunosuppressants (drugs that weaken the immune system) after a transplant to stop the immune system from attacking the new kidney. However, after a kidney transplant fails and patients return to dialysis, there's no clear evidence that continuing immunosuppressants helps prevent allosensitization. Plus, these drugs have serious risks, including infections, heart disease, and even cancer.

The PART study is a pilot study designed to explore whether continuing immunosuppression after a failed transplant for two years (instead of stopping after six months) can lower the risk of allosensitization and whether it is safe to do so. This pilot will also gather data that will be used for a larger trial in the future.

The study will be done at 12 different research centers, and around 96 patients will be enrolled in the pilot trial. The ultimate goal is to better understand if continuing immunosuppressants after transplant failure can make a difference, and whether it's safe enough to proceed to a larger, more definitive trial.

DETAILED DESCRIPTION:
The PART study is designed to evaluate the feasibility and potential benefit of continuing immunosuppressive therapy (IMSN) after kidney transplant failure, specifically to reduce the risk of allosensitization, which complicates the potential for future kidney transplantation. Transplantation remains the preferred treatment for kidney failure but often does not provide a permanent solution, with many transplanted kidneys failing within 12 years. This necessitates either dialysis or a second transplant.

A significant barrier to repeat kidney transplantation is the phenomenon of allosensitization. Allosensitization occurs when the immune system becomes sensitized to foreign human leukocyte antigen (HLA) markers from a failed kidney transplant. This immune response makes it difficult to match patients with subsequent donor kidneys, severely limiting their chances of receiving a second transplant. One of the current practices to mitigate allosensitization involves the continuation of immunosuppressive therapy after kidney transplant failure to reduce immune reactivity to the failed transplant. However, there is insufficient controlled, prospective evidence that this approach is effective in preventing further sensitization or improving outcomes.

Additionally, continuing IMSN after transplant failure carries significant risks, including increased susceptibility to infections, cardiovascular disease, and cancers, all of which contribute to patient morbidity. The current consensus in transplant guidelines recommends discontinuing IMSN after a year post-transplant, yet a multi-center prospective observational study has shown considerable practice variation in Canada, with 65% of patients continuing IMSN beyond the recommended time frame.

This pilot study, which is part of the larger planned PART trial, aims to determine the feasibility of continuing IMSN for two years after transplant failure, compared to withdrawing IMSN at six months. Specifically, the study seeks to demonstrate whether such an intervention can result in a clinically meaningful reduction in allosensitization while maintaining an acceptable level of safety. The findings from this pilot will provide critical data on the feasibility of recruitment, adherence to treatment protocols, and the collection of necessary event outcomes, which will inform the design of a larger, definitive trial.

Study Objectives and Design

The objectives of the PART pilot study are multifaceted. The primary goal is to assess the feasibility of continuing IMSN for two years post-transplant failure. This includes:

Adherence: The study aims to show that more than 80% of enrolled patients adhere to at least 80% of their prescribed IMSN according to the study protocol.

Enrollment: The study aims to demonstrate an enrollment rate of 0.66 patients per month (or 8 patients per 12-month period) across 12 pilot sites, resulting in a total of 96 patients enrolled.

Loss to Follow-up: The goal is to have a loss to follow-up rate of less than 5%, which aligns with rates seen in previous randomized controlled trials (RCTs) involving dialysis patients.

Secondary objectives include validating event outcome rates from prior observational studies to estimate sample size for a definitive trial. These outcomes will include:

Primary efficacy outcome: A clinically significant increase in sensitization, defined by a significant rise in the calculated panel reactive antibody (cPRA) level.

Repeat transplantation rates as a secondary measure of success. Safety outcomes: This includes monitoring for adverse events such as death, new cancer diagnoses, graft intolerance syndrome, hospitalization for infections, and adrenal insufficiency.

Residual renal function: As a potential surrogate marker for dialysis survival, the study will examine if IMSN can help preserve kidney function in patients whose transplant has failed.

The study will be a multi-center, randomized controlled trial with 12 participating centers, and will enroll a total of 96 patients. These patients will be randomized to either continue IMSN for two years or withdraw from IMSN by six months post-dialysis initiation.

Statistical Considerations and Power Analysis

The primary safety endpoints in the study will include critical events such as death, new cancer diagnoses, graft intolerance syndrome, hospitalization for infection, high levels of sensitization (cPRA ≥95%), and adrenal insufficiency. Secondary validating endpoints will include the rate of clinically relevant increases in sensitization, repeat transplantation rates, residual renal function, health-related quality of life, and patient perspectives on IMSN use post-transplant failure.

The statistical analysis will be conducted to ensure robust data collection and analysis for the definitive trial. Each of the 12 pilot sites will randomize 8 patients during the 12-month recruitment period. This provides an overall sample size of 96 patients. The sample size will be sufficient to generate a 95% confidence interval for adherence, assuming a true adherence rate of 80%. These data will be essential in refining the sample size estimates for the definitive PART trial, which will involve approximately 780 patients. The definitive trial will aim for more than 90% power to demonstrate a 30% reduction in sensitization for patients continuing IMSN for two years compared to those withdrawing from IMSN by 180 days after starting dialysis.

Key assumptions for the definitive trial include:

48% of patients stopping IMSN will experience a clinically significant increase in sensitization.

A hazard ratio (HR) of 0.7 for patients continuing IMSN is expected based on prior observational data showing a 40% lower incidence of sensitization in those who continue IMSN compared to those who stop.

Adherence: A target of 80% adherence is anticipated based on pilot trial outcomes.

Repeat transplant rate of 14%, as observed in the prospective observational study.

Death rate of 12% and a loss to follow-up rate of 7%, consistent with findings in previous observational studies.

The data from the PART pilot trial will thus help ensure that the future definitive trial is appropriately designed, with reliable sample size estimates and an accurate understanding of treatment adherence and safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old with a failed first kidney transplant and planned dialysis start date.

Exclusion Criteria:

* Previous extra-renal organ transplant, or more than one previous kidney transplant
* Not prescribed tacrolimus or cyclosporine at the time of transplant failure
* Active infection or cancer that precludes IMSN, or non-transplant indication to continue IMSN
* Receipt of an HLA identical donor transplant kidney with low risk for sensitization
* Patients without archived donor samples to determine eplet mismatch and donor specific antibodies
* Planned nephrectomy of the failed allograft
* Graft survival of ≤ 12 months due to rejection
* Designated as non-repeat transplant candidates by their transplant center or cPRA ≥ 90% at the time of enrollment in whom further increase in cPRA may permanently preclude repeat transplantation
* Planned living donor transplant or planned move away from study center

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
A clinically relevant increase in sensitization | From enrollment to the study at 24 months
  A clinically relevant increase in sensitization defined as an increase in sensitization that decreases the number of HLA compatible donors that a patient can receive a transplant from by at least 50%, is the primary outcome for the future definitive PART Trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Kidney Transplant Research, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No